CLINICAL TRIAL: NCT00517725
Title: Nebivolol Versus Bisoprolol Versus Carvedilol in Heart Failure: Effects on Exercise Capacity and Hypoxia, Chemoreceptor Response, Pulmonary Function
Brief Title: Nebivolol Versus Bisoprolol Versus Carvedilol in Heart Failure
Acronym: CARNEBI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Piergiuseppe Agostoni, Centro Cardiologico Monzino - Univeristy of Milan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R76-CCM S78/407
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Heart Failure
Keywords: exercise; lung diffusion; hypoxia; chemoreceptor; beta-blockers; heart failure
MeSH Terms: conditions — Motor Activity; Hypoxia; Heart Failure | interventions — Carvedilol; Bisoprolol; Nebivolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carvedilol (Active Comparator)
  Interventions: Drug: carvedilol
- Bisoprolol (Active Comparator)
  Interventions: Drug: bisoprolol
- Nebivolol (Active Comparator)
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: carvedilol
  Arms: Carvedilol
Drug: bisoprolol
  Arms: Bisoprolol
Drug: Nebivolol
  Arms: Nebivolol

SUMMARY:
The investigators test the hypothesis that different beta-blockers had a different influence on chemoreceptor response and lung diffusion capacity.

Both could influence exercise capacity in normoxic as well as hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patients in stable clinical condition

Exclusion Criteria:

* No comorbidity
* NYHA class IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
exercise capacity | two months

SECONDARY OUTCOMES:
lung diffusion | two months

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD, PhD, Principal Investigator — Centro Cardiologico Monzino; Giancarlo Marenzi, MD, Study Chair — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, University of Milan, Milan, Italy

REFERENCES:
- [Background] Agostoni P, Bussotti M, Cattadori G, Margutti E, Contini M, Muratori M, Marenzi G, Fiorentini C. Gas diffusion and alveolar-capillary unit in chronic heart failure. Eur Heart J. 2006 Nov;27(21):2538-43. doi: 10.1093/eurheartj/ehl302. Epub 2006 Oct 6. PMID 17028107
- [Derived] Karsten M, Contini M, Cefalu C, Cattadori G, Palermo P, Apostolo A, Bussotti M, Magri D, Salvioni E, Farina S, Sciomer S, Catai AM, Agostoni P. Effects of carvedilol on oxygen uptake and heart rate kinetics in patients with chronic heart failure at simulated altitude. Eur J Prev Cardiol. 2012 Jun;19(3):444-51. doi: 10.1177/1741826711402736. Epub 2011 Mar 7. PMID 21450573